CLINICAL TRIAL: NCT01304719
Title: A Computer-based Intervention to Augment Home Visitation Services: The E-Parenting Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 092506B3F
Record Dates: First submitted 2011-02-10; First posted 2011-02-25 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Child Maltreatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Computer Assisted home visitation (Experimental): Home visitation with computer modules added
  Interventions: Behavioral: Computer Assisted Healthy Families America Home Visitation
- Home Visitation TAU (Experimental): Home Visitation Treatment as Usual
  Interventions: Behavioral: Healthy Families America Home Visitation
- Community Referral (No Intervention): Community Referral

INTERVENTIONS:
Behavioral: Computer Assisted Healthy Families America Home Visitation — Computer modules added to home visitation protocol for Healthy Families America
  Arms: Computer Assisted home visitation
Behavioral: Healthy Families America Home Visitation — Healthy Families America Home Visitation Treatment as Usual
  Arms: Home Visitation TAU

SUMMARY:
The current protocol aims to examine the effects of a computer-based intervention used in conjunction with existing Healthy Families America (HFA) home visitation programs on the challenges related to participant enrollment, retention, and motivation as well as parent and child outcomes.

DETAILED DESCRIPTION:
The present study aims to determine whether a computer-based intervention can provide augmentation of home visiting services to decrease the risk of child maltreatment. The computer-based software includes modules on motivation, Cognitive Retraining, and elements of the ecobehavioral SafeCare approach. A total of 420 mother-infant dyads from four Healthy Families America (HFA) sites will be randomly assigned to either treatment as usual, software-supplemented home visitation, or community control conditions. For families in the software-supplemented condition, home visitors will present the software to parents via a Tablet PC during regular home visits. All parents will be followed-up at 6, 12, and 18 months by independent and blinded research assistants. Parents are evaluated for maltreatment and maltreatment risks as measured by self-report, home visitor report, blinded independent observers, and statewide CPS data. If validated, the proposed intervention can provide augmentation of home visiting services with unprecedented ease of dissemination, at negligible additional cost, and with limitless potential for further development.

ELIGIBILITY:
Inclusion Criteria:

Pregnant or post-partum mothers who are eligible (i.e., score 25 or greater on the Kempe Family Stress Checklist and are not involved in CPS open case investigation at the time of HFA participation) and willing to participate in the HFA program are eligible to participate in the current study, with the following restrictions:

1. Mothers must be 18 years or older and able to complete the baseline assessment within 4 weeks of delivery.
2. Mothers have not completed any prior post-partum treatment plan.
3. Participants must have functional cognitive abilities.
4. Premature infants have to be released from hospital care within 6 weeks of birth.
5. Participants must be able to communicate in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Child maltreatment reports | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Ondersma, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States